CLINICAL TRIAL: NCT04296929
Title: The Effect of Complex Decongestive Physiotherapy on Sensory Parameters in Breast Cancer Related Lymphedema Patients
Brief Title: The Effect of Complex Decongestive Physiotherapy on Sensory Parameters in Breast Cancer Related Lymphedema.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine BARAN, Research Assistant, Physical Therapist, Master of Science, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBaran
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Lymphedema; Lymphedema of Upper Arm; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affected arm in lymphedema patients (Experimental): Complex decongestive physiotherapy treatment will be applied to the arm (affected arm) that develops lymphedema after unilateral breast cancer treatment.
  Interventions: Other: Complex Decongestive Physiotherapy
- Unaffected arm in lymphedema patients (No Intervention): After unilateral breast cancer treatments, the non-lymphedema side in the upper extremities, is the unaffected arm. No treatments will be applied to the unaffected side.

INTERVENTIONS:
Other: Complex Decongestive Physiotherapy — Complete decongestive therapy (CDT), also called complex decongestive therapy, is an intensive program that combines many of the different treatment approaches, including bandaging, compression garments, manual lymphatic drainage, exercise, and self care.
  Arms: Affected arm in lymphedema patients

SUMMARY:
The aim of this study was to determine the effect of complex decongestive physiotherapy in women with unilateral breast cancer-related lymphedema on sensory parameters.

DETAILED DESCRIPTION:
Although there are a limited number of studies in the literature on disorders of sensory functions seen after breast cancer treatments, sensory disorders that may be seen in lymphedema associated with breast cancer were evaluated in only 2 studies published in 1979 and 2006. Although these studies are not sufficient in terms of study design, they only include Semmes-Weinstein monofilaments and two-point discrimination tests and hand evaluations. Ganel et al. Reported that approximately 50% of the patients they included in the study found that varying degrees of lymphedema developed in the upper extremity, and the median nerve compression in the brachial plexus and carpal tunnel was significantly higher in these patients. They did not find a direct correlation with radiotherapy in patients with nerve compression. They therefore stated that nerve compression may be associated with lymphedema or fibroblast infiltration. According to this study, lymphedema may also be a risk factor in post mastectomy problems such as brachial plexus and carpal tunnel syndrome. Greve et al. reported that lymphedema may cause a decrease in sensory functions in patients who were evaluated with monofilaments in their studies on the effect of lymphedema on sensory functions after mastectomy (Ganel 1979, Greeve 2006).

Complex Decongestive Physiotherapy was developed by Földi in the 1980s in Germany to reduce limb volume, preserve skin health, lymph transport stimulation and reabsorption of residual interstitial proteins. Complex Decongestive Physiotherapy is a treatment method consisting of four main elements and two phases. The four main elements of the first phase of complex decongestive physiotherapy; includes manual lymphatic drainage, skin care, compression therapy and remedial exercises. After the edema is reduced, phase II is passed. This phase includes self-drainage, skin care, personalized compression socks and remedial exercises. In lymphedema, protein-rich fluid accumulates in the subcutaneous tissue for a long time, disrupting natural skin elasticity over time. With Complex Decongestive Physiotherapy, edema reduction up to 65% can be achieved, functional loss, fibrotic changes, and cosmetic problems, which are the secondary problems caused by lymphedema, can be observed.

Increased interstitial fluid in lymphedema associated with breast cancer can cause local sensory loss due to compression of peripheral nerves. Dermal thickness increase due to lymphedema and biomechanical changes in viscoelasticity can cause various changes on sensory functions. Therefore, quantitative evaluation of the sensory system can be an effective method to determine the injury risk factor of the lymphedema region in the event of an existing sensory dysfunction. However, although the effects of Complex Decongestive Physiotherapy on edema reduction, skin thickness and elasticity are mentioned, its effect on sensory functions is unknown.

Complex Decongestive Physiotherapy will be applied to patients for a total of 3 weeks, 5 days a week within the scope of this study.

The assessments will be performed before treatment and at the end of three weeks treatment period.

A detailed story will be taken from the patients first. The lymphedema diagnoses of the patients will be confirmed by ultrasonographic imaging method. Imaging will be performed using a 5-12 MHz linear probe (Logiq P5, GE, Wisconsin, USA) on the upper extremity. Dermis and subcutaneous soft tissue thicknesses; It will be measured using plenty of gel, using images without applying any pressure - with the help of the device's automatic calculation feature after marking.

The severity of lymphedema between the two extremities will be assessed by environmental measurement.

Semmes-Weinstein Monofilament Test: It will be applied 10 cm distal to the elbow joint of the volar surface in the forearm. The measurement will start with the lightest monofilament and proceed to the monofilament that the patient feels. Each monofilament will be applied to a spot three times in a row.

Two Point Discrimination Test: This test is a non-invasive test commonly used in sensory evaluation. It is done by randomly touching one or two points. If 7 of the 10 answers given by the patient are correct, the answer is considered correct. If the answer is not correct, the difference between the two ends of the esthesiometer is increased by 1, 2 or 5 mm depending on the expected state of sensory loss. The test continues until you reach the correct answer. If the correct answer cannot be obtained even at 15 mm, the test is terminated.

The pressure pain threshold will be evaluated with 'J tech Algometer Commander' by giving pressure from both the upper extremity to 10 cm distal from the volar surface of the elbow joint until the patient feels minimal pain. Pressure will be applied vertically with the 1 cm2 head of the device and patients will be asked to say 'yes' whenever they feel uncomfortable with the pressure applied. The measurement will be repeated 3 times, and the pressure pain threshold will be calculated by taking the arithmetic average of these three trials.

Hot / Cold Sensory Test: The sense of warm / cold will be evaluated with test tubes containing hot and cold liquid. The cold tube will be filled with water at 10 °C and the hot tube at 40 °C. When the patient's eyes are closed, these tubes will be touched to the skin surface 10 cm distal to the volar face elbow joint in a random order, and the patient will be asked to express that the water in the tube is hot or cold.

Vibration Sensation Measurement: The vibration sensation will be measured from the lateral epicondyle in the upper extremity by diapason. Diapason is a small U-shaped tool made of steel that vibrates at a certain height when vibrated.

Lymphedema Life Impact Scale: Weiss et al. The validity and reliability of the questionnaire developed by Orhan et al. made by. Lymphedema life impact scale consists of 18 questions and has physical, psychological and functional subtitles. '0'; no influence, '4'; It is scored between the minimum '0' and the maximum '72' score with a 5-stage Likert-type scale in the form of severe influence. As the score increases, the state of influence worsens.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lymphedema disease
* Ages between 18-80 years old,
* 2 cm difference between the affected and unaffected arms in women with breast cancer related lymphedema,
* At least 12 months after breast cancer treatments end and
* Who are agreed to participate in the study.

Exclusion Criteria:

* Women with active infection,
* deep vein thrombosis/thrombophlebitis,
* cardiac edema,
* peripheral artery disease,
* kidney, lung disease,
* primary lymphedema,
* peripheral upper limb nerve injury,
* any surgery other than breast cancer surgeries,
* existing shoulder, elbow, wrist, hand pathologies,
* cooperation problems,
* neurological disease,
* mental illness, diabetes mellitus,
* smoking and patients with open wounds on the upper limb.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was planned in women with breast cancer related lymphedema.
Enrollment: 30 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Touching sensation | Change from Baseline touching sensation at 3 weeks
  Assessment of touching sensation at 10 cm distal to the elbow on the volar surface in affected and unaffected arms at least 12 months after the breast cancer treatment, with Semmes-Weinstein Monofilaments in women with breast cancer related lymphedema.
Two-point discrimination | Change from baseline two-point discrimination at 3 weeks
  Assessment of two-point discrimination at 10 cm distal to the elbow on the volar surface in affected and unaffected arms at least 12 months after the breast cancer treatment, with an esthesiometer in women with breast cancer related lymphedema.
Pressure pain threshold | Change from baseline pressure pain threshold at 3 weeks
  Assessment of pressure pain threshold at 10 cm distal to the elbow on the volar surface in affected and unaffected arms at least 12 months after the breast cancer treatment, with an algometer in women with breast cancer related lymphedema.

SECONDARY OUTCOMES:
Vibration sensation | Change from baseline vibration sensation at 3 weeks
  Vibration Sensation Measurement: The vibration sensation will be measured from the lateral epicondyle in the upper extremity by diapasons. Diapason is a small U-shaped tool made of steel that vibrates at a certain height when vibrated. 128 and 256 Hertz diapasons will be vibrated and placed in the patient's lateral epicondyle. The time that the patient feels vibration will be calculated with a chronometer.
Ultrasonographic Imaging | Change from baseline ultrasonographic imaging at 3 weeks.
  The lymphedema diagnoses of the patients will be confirmed by ultrasonographic imaging method routinely performed in the clinic. Imaging will be performed using a 5-12 MHz linear probe (Logiq P5, GE, Wisconsin, USA) on the upper extremity. Dermis and subcutaneous soft tissue thicknesses; It will be measured using plenty of gel, using images without applying any pressure - with the help of the device's automatic calculation feature after marking.
Environmental measurement | Change from baseline environmental measurement at 3 weeks.
  The severity of lymphedema between the two extremities will be measured by measuring the environment at 5 cm intervals.
Hot / Cold Sensory Test | Change from baseline Hot/Cold sensory Test at 3 weeks
  The sense of warm / cold will be evaluated with test tubes containing hot and cold liquid. The cold tube will be filled with water at 10 ° C and the hot tube at 40 ° C. When the patient's eyes are closed, these tubes will be touched to the skin surface 10 cm distal to the volar face elbow joint in a random order, and the patient will be asked to express that the water in the tube is hot or cold.
Lymphedema Life Impact Scale | Change from baseline Lymphedema Life Impact Scale at 3 weeks.
  Lymphedema Life Impact Scale: Weiss et al. The validity and reliability of the questionnaire developed by Orhan et al. made by. Lymphedema life impact scale consists of 18 questions and has physical, psychological and functional subtitles. '0'; no influence, '4'; It is scored between the minimum '0' and the maximum '72' score with a 5-stage Likert-type scale in the form of severe influence. As the score increases, the state of influence worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Ribeiro Pereira ACP, Koifman RJ, Bergmann A. Incidence and risk factors of lymphedema after breast cancer treatment: 10 years of follow-up. Breast. 2017 Dec;36:67-73. doi: 10.1016/j.breast.2017.09.006. Epub 2017 Oct 6. PMID 28992556
- [Background] Rijke AM, Croft BY, Johnson RA, de Jongste AB, Camps JA. Lymphoscintigraphy and lymphedema of the lower extremities. J Nucl Med. 1990 Jun;31(6):990-8. PMID 2348245
- [Background] Goyal A, Newcombe RG, Chhabra A, Mansel RE. Morbidity in breast cancer patients with sentinel node metastases undergoing delayed axillary lymph node dissection (ALND) compared with immediate ALND. Ann Surg Oncol. 2008 Jan;15(1):262-7. doi: 10.1245/s10434-007-9593-3. Epub 2007 Sep 19. PMID 17879117
- [Background] Wu SG, Huang SJ, Zhou J, Sun JY, Guo H, Li FY, Lin Q, Lin HX, He ZY. Dosimetric analysis of the brachial plexus among patients with breast cancer treated with post-mastectomy radiotherapy to the ipsilateral supraclavicular area: report of 3 cases of radiation-induced brachial plexus neuropathy. Radiat Oncol. 2014 Dec 12;9:292. doi: 10.1186/s13014-014-0292-5. PMID 25499205
- [Background] Warmuth MA, Bowen G, Prosnitz LR, Chu L, Broadwater G, Peterson B, Leight G, Winer EP. Complications of axillary lymph node dissection for carcinoma of the breast: a report based on a patient survey. Cancer. 1998 Oct 1;83(7):1362-8. doi: 10.1002/(sici)1097-0142(19981001)83:73.0.co;2-2. PMID 9762937
- [Background] Andersen KG, Duriaud HM, Kehlet H, Aasvang EK. The Relationship Between Sensory Loss and Persistent Pain 1 Year After Breast Cancer Surgery. J Pain. 2017 Sep;18(9):1129-1138. doi: 10.1016/j.jpain.2017.05.002. Epub 2017 May 11. PMID 28502878
- [Background] Say CC, Donegan W. A biostatistical evaluation of complications from mastectomy. Surg Gynecol Obstet. 1974 Mar;138(3):370-6. No abstract available. PMID 4811322
- [Background] Ganel A, Engel J, Sela M, Brooks M. Nerve entrapments associated with postmastectomy lymphedema. Cancer. 1979 Dec;44(6):2254-9. doi: 10.1002/1097-0142(197912)44:63.0.co;2-9. PMID 509395
- [Background] Foldi M, Foldi E. [Therapy of lymphedema]. Med Welt. 1980 May 23;31(21):801-6. No abstract available. German. PMID 6993841
- [Background] Lim CY, Seo HG, Kim K, Chung SG, Seo KS. Measurement of lymphedema using ultrasonography with the compression method. Lymphology. 2011 Jun;44(2):72-81. PMID 21949976
- [Background] Voerman VF, van Egmond J, Crul BJ. Normal values for sensory thresholds in the cervical dermatomes: a critical note on the use of Semmes-Weinstein monofilaments. Am J Phys Med Rehabil. 1999 Jan-Feb;78(1):24-9. doi: 10.1097/00002060-199901000-00007. PMID 9923425
- [Background] MOBERG E. Objective methods for determining the functional value of sensibility in the hand. J Bone Joint Surg Br. 1958 Aug;40-B(3):454-76. doi: 10.1302/0301-620X.40B3.454. No abstract available. PMID 13575459
- [Background] Dellon AL. The moving two-point discrimination test: clinical evaluation of the quickly adapting fiber/receptor system. J Hand Surg Am. 1978 Sep;3(5):474-81. doi: 10.1016/s0363-5023(78)80143-9. PMID 568154
- [Background] Granges G, Littlejohn G. Pressure pain threshold in pain-free subjects, in patients with chronic regional pain syndromes, and in patients with fibromyalgia syndrome. Arthritis Rheum. 1993 May;36(5):642-6. doi: 10.1002/art.1780360510. PMID 8489541
- [Background] Weiss J, Daniel T. VALIDATION OF THE LYMPHEDEMA LIFE IMPACT SCALE (LLIS): A CONDITION-SPECIFIC MEASUREMENT TOOL FOR PERSONS WITH LYMPHEDEMA. Lymphology. 2015 Sep;48(3):128-38. PMID 26939160
- [Background] Orhan C, Uzelpasaci E, Baran E, Nakip G, Ozgul S, Aksoy S, Akbayrak T. The Reliability and Validity of the Turkish Version of the Lymphedema Life Impact Scale in Patients With Breast Cancer-Related Lymphedema. Cancer Nurs. 2020 Sep/Oct;43(5):375-383. doi: 10.1097/NCC.0000000000000709. PMID 30921030
- [Derived] Baran E, Ozcakar L, Ozgul S, Aksoy S, Akbayrak T. Upper limb sensory evaluations and ultrasonographic skin measurements in breast cancer-related lymphedema receiving complex decongestive physiotherapy. Support Care Cancer. 2021 Nov;29(11):6545-6553. doi: 10.1007/s00520-021-06235-4. Epub 2021 Apr 29. PMID 33913006